CLINICAL TRIAL: NCT04346212
Title: Oropharyngeal Dysphagia and Malnutrition in Patients Infected by SARS-CoV-2: Prevalence and Needs of Compensatory Treatment and Follow up in Patients Admitted by COVID-19 at the Consorci Sanitari Del Maresme
Brief Title: Oropharyngeal Dysphagia in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital de Mataró (Other)
Collaborators: Centro Investigación Biomédica en Red de Enfermedades Hepáticas Digestivas (Unknown)
Responsible Party: Principal Investigator, Pere Clave, Director of Research and Academic Development at CSdM, Hospital de Mataró
Other Study IDs: COVID_OD
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Oropharyngeal Dysphagia; COVID-19; Sars-CoV2; Nutrition
MeSH Terms: conditions — Deglutition Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients infected by SARS-CoV-2: Patients infected by SARS-CoV-2 at the Hospital de Mataró, Hospital de St. Jaume i Sta. Magdalena and other medicalized facilities in Mataró.
  Interventions: Diagnostic Test: Swallowing evaluation with the EAT-10 and the volume-viscosity swallowing test (V-VST)

INTERVENTIONS:
Diagnostic Test: Swallowing evaluation with the EAT-10 and the volume-viscosity swallowing test (V-VST) — We will assess dysphagia, nutritional status and needs of compensatory treatment (fluid and nutritional adaptation) in patients with COVID-19 disease. We will also collect clinical data, information about swallowing and nutritional status and needs through the electronical medical history of the patients and by telephone call at 3 and 6 months follow-up, as well as clinical complications.
  Other Names: Nutritional evaluation (NRS 2002); Fluid and nutritional adaptation registry (needs of compensatory treatment); Clinical complications at 6 months

SUMMARY:
Background: Oropharyngeal dysphagia (OD) is a common complication in/post ICU patients that have been with intubation/mechanical ventilation or with tracheotomies or NG tubes, in patients with acute respiratory infection/pneumonia/respiratory insufficiency with a severe disease needing high concentration of oxygen or noninvasive mechanical ventilation and also in patients discharged from acute hospitals to rehabilitation centers, nursing homes or other facilities. All these situations are common for COVID-19 patients that are currently filling our hospitals due to the pandemic expansion of SARS-CoV-2. OD is associated to prolonged hospitalization, dehydration and severe nutritional and respiratory complications -aspiration pneumonia-, hospital readmissions and mortality. Aim: to assess the prevalence of OD and nutritional risk in these patients and to know their needs of compensatory treatment following the application of an early intervention, and to assess whether OD and malnutrition are indicators of poor prognosis for COVID-19 patients. Methods: prospective study in which we will use the volume-viscosity swallowing test (V-VST) to assess the prevalence of OD, and NRS2002 to assess the nutritional risk in admitted patients with confirmed COVID-19 at the Consorci Sanitari del Maresme, Catalonia, Spain. We will register also results of the EAT-10, nutritional status, the needs of compensatory treatments of these patients following an early intervention with fluid and nutritional adaptation and use of nutritional supplements. We will also collect other clinical variables from medical history of the patient related to hospitalization and we will follow the clinical complications and nutritional status at 3 and 6 months follow up.

DETAILED DESCRIPTION:
Design: 1) prospective study in SARS-CoV-2 infected patients admitted to the CSdM more than 48h with 2 follow-up points at 3/6 months after discharge.

2) comparative study between the 3 first waves of the pandemic in the acute phase.

Aims:

1.1)To assess the prevalence of OD, nutritional risk, the needs of compensatory treatment and complications at 3/6 month follow up of patients admitted by COVID-19 in Hospital de Mataró, Hospital St. Jaume and the medicalized Atenea Hotel, Mataró (Barcelona), Spain.

1.2)To validate an early intervention including fluid thickening and nutritional support.

1.3)In addition, we would like to know if those patients with OD and those with OD and MN have worse prognosis than those without these conditions.

2.1) To compare the three first waves of the pandemic in the hospitalization period (clinical, swallowing, nutritional status and mortality).

* Inclusion criteria: Infected patients (COVID-19 + PCR or according to physician's criteria at discharge medical report) admitted to the CSdM >48h; patients able to be explored regarding OD and nutritional status according to their physician's criteria (fully awake patients in a stable respiratory situation and optimal PaO2/FiO2).
* Exclusion criteria: uncontrolled risk of infection for healthcare professionals (HCP).

Study population

All COVID-19 patients admitted to the CSdM more than 48h from April to the end of the pandemic:

1. ICU. Patients in/post ICU with OD associated with intubation/mechanical ventilation or OD associated with tracheotomies or NG tubes (semi-critical patients).
2. Wards. Patients with respiratory infection/pneumonia/respiratory insufficiency, some of them with a severe disease needing high concentration of oxygen or noninvasive mechanical ventilation (acute patients with some complexity).
3. Post-acute COVID-19 patients discharged from acute hospitals to rehabilitation centers, nursing homes or medicalized facilities (sub-acute patients, convalescents).

Sample size calculation: Taking into account the main study variable and that we will do an opportunistic recruitment (admitted patients), a sample size of 315 subjects randomly selected will suffice to estimate with a 95% confidence and a precision +/-5.5 percent units, a population percentage considered to be around 55.0% (estimated OD prevalence). It has been anticipated a replacement rate of 0%.

Study variables

* Main variable: prevalence of OD and risk of malnutrition among COVID-19 patients.
* Secondary variables: needs of nutritional supplementation, texture-modified diets, use of thickeners and patient's adherence to compensatory measures, functional capacity, comorbidities, nutritional analytical parameters, weight, clinical severity (including pneumonia severity), neurological symptoms, pharmacological treatment, ICU admission, and hospital readmissions, visits to emergency department, respiratory infections and mortality at 3 and 6 months follow-up. Clinical prognosis in those patients with OD and/or MN compared to those without these conditions.

Study visits/evaluations/management 4 evaluation points*: 1) admission; 2) discharge; and 3-4) follow up at 3 months and 6 months. According to the first evaluation, an interventional plan (management) will be prescribed in order to improve patient's swallowing, feeding and nutritional status during admission. All the evaluations and interventional plans are currently being performed as standard clinical practice and will be obtained from patient's medical history record. Study variables will be grouped in 3 different assessments: a) clinical assessment; b) swallowing assessment; and c) nutritional assessment.

* There will be no follow-up in the comparative study between the 3 firsts waves of the pandemic.

1. Admission*: there will be 2 admission evaluation points, the first one 24-48h after admission (pre-admission data) and the second one during admission (admission data).

   1.1.Clinical evaluation: patient origin (community, nursing home, socio-health center), functional status before, during admission and at discharge (Barthel index), comorbidities (Charlson index), clinical symptoms before and during admission, neurological symptoms, ICU admission and length of stay, respiratory infection, its symptoms, severity and length from the week before admission, prescribed pharmacological treatment, hospitalization days and mortality during admission.

   1.2.Swallowing evaluation: anamnesis, EAT-10 questionnaire (screening), clinical swallowing assessment with volume-viscosity swallowing test (V-VST) at admission and tolerance and adherence with the recommendations (volume and viscosity) during admission.

   1.3.Nutritional evaluation: anthropometrical measurements and nutrition-related questions pre and post-admission, analytical parameters at admission and during admission (albumin, pre-albumin, cholesterol, total proteins, lymphocytes, ferritin and C-reactive protein), NRS2002 at admission and at discharge and nutritional recommendations during admission (ONS, type of diet and intake) and patient's adherence.
2. Discharge:

   2.1.Codification at discharge: SARS-CoV2 pneumonia, OD, respiratory infection, aspiration pneumonia, malnutrition or others.

   2.2.Recommendations at discharge: fluid and nutritional recommendations at discharge (volume and viscosity, oral nutritional supplementation and type of diet).

   *After evaluations, healthcare professionals will give to the patients clinical recommendations on the use of thickeners, texture-modified diets and nutritional supplementation if required.
3. Follow up (3/6 months): we will collect clinical data, information about swallowing and nutritional status and needs through the electronical medical history of the patients and by telephone call. Patients will receive new recommendations on fluid and nutritional adaptation and nutritional supplementation if required. The follow-up evaluations will include:

3.1.Clinical evaluation: mortality (date), patient residence (community, nursing home, socio-health center), functional status (Barthel index), and hospital resources consumption/clinical outcomes (hospital readmissions, visits to the emergency department, and respiratory infections).

3.2.Swallowing evaluation: anamnesis, EAT-10 (swallowing screening); if positive, virtual clinical swallowing assessment with the V-VST, and fluid adaptation recommendations.

3.3.Nutritional evaluation: anthropometrical measurements (current weight), ONS intake (time taken from discharge), textural diet adaptation if needed and compliance with the previous recommendations, NRS2002, and analytical parameters (albumin, cholesterol, ferritin, C-reactive protein) if the patient had a blood analysis during the previous month.

Management of patients with COVID-19, OD and MN:

After admission in our health care centers, COVID-19 patients will be screened by a speech and language pathologist (SLP) for OD with specific questions and the V-VST, and nutritional status with the NRS2002. In addition, clinical data of patients will be recorded during admission. Those patients with a NRS2002 ≥ 3 points, will require ONS, that will be given in two formats (liquid or viscosity-adapted) depending on the swallowing status. Those patients with less than 70 years will receive 2 instead of 1/day. According to patient's masticatory and swallowing hability they will receive texture-modified diets in 3 different formats: 1) normal, 2) easy mastication diet, and 3) puree. Normal diet is composed by 1750Kcal/70g protein; if the patient is at nutritional risk or malnourished (NRS2002≥3) he/she will also receive a high caloric-proteic diet with 2000Kcal/90g protein. Finally there will be a fluid adaptation according to the results of the V-VST with 3 different viscosities: 1)liquid, 2)250mPa•s, and 3)800mPa•s. During admission patients will be managed by the SLPs and the nutritionist team of the healthcare centers. Just before discharge, patients will be re-evaluated and swallowing and nutritional recommendations will be given adapted to the new status of the patient by using the same criteria. On a nutritional level, just before discharge, patients will be re-evaluated by the team of dietitians to detect those patients who have not yet improved their nutritional status and therefore will need to continue taking ONS after discharge. The criteria for maintaining or not maintaining the prescription at discharge will be those corresponding to a normal dietary assessment, such as: anorexia, not having recovered weight or insufficient intake due to vomiting, nausea or other causes not related to hospital food. Other criteria may be included at the discretion of the clinical professional. This group will be dispensed ONS for at least 1 month after discharge.

We will collect also data on patient's destination, functional capacity, weight loss, admission to the ICU and clinical data at discharge. Finally, patients will be followed-up at 3/6 months for clinical complications through their electronic medical history.

Main study procedures and variables

* EAT-10: is a simple 10-item questionnaire to screen for the risk of dysphagia (score>2, risk of OD) (Belafsky P 2008, Ann Otol Rhinol Laryngol; Rofes L 2014, Neurogastroenterol Motil).
* V-VST: is a validated clinical test to explore safety and efficacy of swallow and select the optimal bolus volume and viscosity for each patient with/at risk of OD. It uses different volumes (5, 10 and 20mL) and viscosities (250mPa•s, liquid and 800mPa•s) (thickener Nutilis Clear) to evaluate clinical signs of impaired efficacy and safety of swallow. We will apply a simplified V-VST with only 1 volume (10mL) and the 3 usual viscosities in order to reduce the hospital burden and stress for the patient (Clavé P 2008, Clin Nutr). Recommendations on fluid adaptation given to the patient according to the results of the test will be recorded.
* Nutritional status: a nutritional evaluation is done to COVID-19 patients according to their phenotype. We will use the nutritional risk screening (NRS 2002), a validated nutritional screening tool for hospitalized adult patients and has been recommended by a recent guideline for COVID-19 admitted patients (Ying-Hui Jin, 2020, Mil Med Res). If the patient scores 3 or more points is considered to be in nutritional risk and a more comprehensive nutritional evaluation should be performed and nutritional supplementation applied. Recommendations on nutritional adaptation given to the patient (adaptation of texture/calories/proteins and nutritional supplementation) according to the results of the tests will be recorded.
* Other study variables collected from patient's medical history: patient origin and destination at discharge, hospitalization days, admission to the ICU, myopathy post-ICU and length of stay in the ICU, symptomatology before and during admission (fever, cough, dyspnea, diarrhea, vomiting, ageusia, anosmia, headache, polymyalgia), neurological symptoms during admission (seizures, encephalitis, delirium, headache, dyskinesia, stroke, parenthesis, ataxia, encephalitis), functionality with the Barthel index (pre-admission, admission and discharge), comorbidities with the Charlson score, respiratory infections during admission and its severity and type, use of oxygen therapy, pronation, prescribed treatment, anthropometric measurements (weight at discharge, weight loss), use and tolerability of oral nutritional supplements, nutritional intake, use of enteral or parenteral nutrition, biochemical parameters at admission and discharge (pre-albumin, albumin, cholesterol, total proteins, lymphocytes, ferritin and C-reactive protein), diagnostics at discharge (SARS-CoV2 pneumonia, OD, respiratory infection, aspiration pneumonia, malnutrition or others), and intra-hospital mortality.
* Follow-up (3 and 6 months): we will collect data of clinical complications from the medical history of the patient and by telephone call: swallowing, nutritional status and needs (including analytical parameters), hospital readmissions, visits to the emergency department, incidence of respiratory infections (including pneumonia, COPD exacerbations) and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Infected patients (COVID-19 + by PCR or according to physician's criteria in the medical report of the patient at discharge) admitted to the CSdM more than 48 h.
* Patients able to be explored regarding OD and nutritional status according to their physician's criteria (fully awake patients in a stable respiratory situation and optimal PaO2/FiO2).

Exclusion Criteria:

* Uncontrolled risk of infection for healthcare professionals (HCP) (according to the safety considerations stated below).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All COVID-19 + patients admitted to the CSdM more than 48h from April to the end of the pandemic (estimation: N=300).
  There are 3 main phenotypes of patients with OD related to COVID-19:
  1. ICU. Patients in/post ICU with OD associated with intubation/mechanical ventilation or OD associated with tracheotomies or NG tubes (critical or semi-critical patients).
  2. Wards. Patients with respiratory infection/pneumonia/respiratory insufficiency, some of them with a severe disease needing high concentration of oxygen or noninvasive mechanical ventilation (acute patients with some complexity).
  3. Post-acute COVID-19 patients discharged from acute hospitals to rehabilitation centers, nursing homes or medicalized facilities (sub-acute patients, convalescents).
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in the prevalence of oropharyngeal dysphagia | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the prevalence of oropharyngeal dysphagia according to a clinical assessment tool, the Volume-Viscosity Swallowing Test (V-VST).

SECONDARY OUTCOMES:
Changes in the swallowing screening | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the eating assessment tool (EAT-10 score). A tool that goes from 0 to 40 points and indicates that the patient is at risk of oropharyngeal dysphagia if he/she presents 3 or more points
Changes in the swallowing status | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the percentage of patients with impairements in efficacy and/or safety of swallow.
Changes in the nutritonal status of study patient's. | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the nutritional status of study patients (% malnourished, at risk of malnutrition or wellnourished).
Changes in the needs of compensatory treatments in those patients with oropharyngeal dysphagia (fluid adaptation). | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the fluid (volume and viscosity) requirements of study patients.
Changes in the needs of compensatory treatments in those patients with oropharyngeal dysphagia (nutritional adaptation). | From April 2020 to September 2021. And at 3 and 6 months follow-up (1st wave).
  Changes in the nutritional adaptation requirements (type of diet and need of nutritional supplementation).
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (incidence of readmissions). | 3 and 6 months from inclusion.
  Changes in the incidence of hospital readmissions: number of hospital readmissions/patient/6 months.
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (prevalence of readmissions). | 3 and 6 months from inclusion.
  Changes in the prevalence: % of patients with hospital readmissions during the follow-up.
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (number of visits to emergency department). | 3 and 6 months from inclusion.
  Incidence: number of visits to the emergency department/patient/ 3 or 6 months.
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (percentage of visits to emergency department). | 3 and 6 months from inclusion.
  Prevalence: % of patients visiting the emergency department during the follow-up.
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (respiratory complications). | 3 and 6 months from inclusion.
  Incidence of respiratory infections (including pneumonia, and COPD exacerbations).
Changes in the clinical complications at 3 and 6 months follow up from patient's medical history (mortality). | 3 and 6 months from inclusion.
  3 and 6 months mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Consorci Sanitari del Maresme (Hospital de Mataró), Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clave P, Shaker R. Dysphagia: current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):259-70. doi: 10.1038/nrgastro.2015.49. Epub 2015 Apr 7. PMID 25850008
- [Background] Ortega O, Martin A, Clave P. Diagnosis and Management of Oropharyngeal Dysphagia Among Older Persons, State of the Art. J Am Med Dir Assoc. 2017 Jul 1;18(7):576-582. doi: 10.1016/j.jamda.2017.02.015. Epub 2017 Apr 12. PMID 28412164
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Background] Rofes L, Arreola V, Mukherjee R, Clave P. Sensitivity and specificity of the Eating Assessment Tool and the Volume-Viscosity Swallow Test for clinical evaluation of oropharyngeal dysphagia. Neurogastroenterol Motil. 2014 Sep;26(9):1256-65. doi: 10.1111/nmo.12382. Epub 2014 Jun 9. PMID 24909661
- [Background] Clave P, Arreola V, Romea M, Medina L, Palomera E, Serra-Prat M. Accuracy of the volume-viscosity swallow test for clinical screening of oropharyngeal dysphagia and aspiration. Clin Nutr. 2008 Dec;27(6):806-15. doi: 10.1016/j.clnu.2008.06.011. Epub 2008 Sep 11. PMID 18789561
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Todorovic V. Detecting and managing undernutrition of older people in the community. Br J Community Nurs. 2001 Feb;6(2):54-60. doi: 10.12968/bjcn.2001.6.2.54. PMID 11927872
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Derived] Martin-Martinez A, Ortega O, Vinas P, Arreola V, Nascimento W, Costa A, Riera SA, Alarcon C, Clave P. COVID-19 is associated with oropharyngeal dysphagia and malnutrition in hospitalized patients during the spring 2020 wave of the pandemic. Clin Nutr. 2022 Dec;41(12):2996-3006. doi: 10.1016/j.clnu.2021.06.010. Epub 2021 Jun 15. PMID 34187698